CLINICAL TRIAL: NCT03986359
Title: Treatment of Erectile Dysfunction With Low-intensity Extracorporeal Shockwave Therapy: A Prospective, Randomized, Single-blind, Cross-over Study
Brief Title: Treatment of Erectile Dysfunction With Low-intensity Extracorporeal Shockwave Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University (Other)
Responsible Party: Principal Investigator, Fu-Shun Hsu, Principal Investigator, National Taiwan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: T-NTUH-57401
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Erectile Dysfunction Following Radiation Therapy
Keywords: low-intensity extracorporeal shockwave therapy; Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: We prospectively assessed the clinical outcome of LI-ESWT for the treatment of ED of organic origin. This study was approved by the institutional review board at National Taiwan University Hospital (NTUH, No. T-NTUH-57401).
Who Masked: Participant
Masking Description: While subjects receive Sham therapy, the machine turning on but the energy is zero.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): 30 subjects receive ESWT (LM-IASO, Litemed Co., Taiwan) for 6 courses in 3 weeks (0.05mJ/mm2, 3000 pulses). Thereafter, the two groups are cross over.
  Interventions: Device: low energy extracorporeal shockwave therapy
- 2 (Sham Comparator): 30 subjects receive Sham therapy for 3 weeks (the machine turning on but the energy is zero). Thereafter, the two groups are cross over.
  Interventions: Device: low energy extracorporeal shockwave therapy

INTERVENTIONS:
Device: low energy extracorporeal shockwave therapy — Low-intensity extracorporeal shockwave therapy (LI-ESWT) was proved to be useful in various medical conditions; for example, neovascularization in myocardial ischemia, nonhealing wounds, ED and chronic pelvic pain syndrome

SUMMARY:
This study is a prospective, randomized, single-blinded, cross-over trial to investigate the efficacy of low-intensity extracorporeal shockwave therapy in the treatment of erectile dysfunction (ED). We will enroll 60 subjects (International Index of Erectile Function Questionnaires, 5 ≦ IIEF-5 ≦ 21). 30 subjects receive ESWT (LM-IASO, Litemed Co., Taiwan) for 6 courses in 3 weeks (0.05mJ/mm2, 3000 pulses) and 30 subjects receive Sham therapy for 3 weeks (the machine turning on but the energy is zero). After 3 weeks, the two groups are cross over. The primary outcome is the 4th week change from baseline for IIEF-5 score. Secondary outcomes are the 8th week change from baseline for IIEF-5 score, EHS, QoL; AEs. The between-group relationships of baseline and 4-week data were evaluated by using the Student's t-test or Mann-Whitney U-test where appropriate. Multiple linear regression was carried out to test the variables associated with treatment outcome. P-values < 0.05 were considered statistically significant.

DETAILED DESCRIPTION:
Low-intensity extracorporeal shockwave therapy (LI-ESWT) was proved to be useful in various medical conditions; for example, neovascularization in myocardial ischemia, nonhealing wounds, ED and chronic pelvic pain syndrome.

The use of LI-ESWT has been increasingly proposed as a treatment for ED over the last decade. Overall, most of these studies reported encouraging results, regardless of variation in LI-ESWT set-up parameters or treatment protocols. As a whole these studies suggest that LI-ESWT could significantly improve the IIEF-5 and Erection Hardness Score of mild ED patients. However, no randomized control trial with cross-over designed studies so far.

This is a prospective, randomized, single-blind, cross-over clinical study. This study will be performed in outpatient setting of NTUH. Written informed consent will be given by all participants before entering the study. The subjects are treated at the therapy room of the department of urology, NTUH. All subjects would not pay any cost for this treatment/study. This study was approved by the institutional review board at National Taiwan University Hospital (NTUH, No. T-NTUH-57401).

Inclusion criteria: were patient age 20 ~ 70 year-old man, suffering from ED for over 6 months, and 5 ≦ IIEF-5 ≦ 21. The written informed consent forms from all subjects who met the inclusion criteria were obtained.

Exclusion criteria: Patients with penile implant, prior radical prostatectomy, rectal surgery, radiation therapy to the pelvic area, spinal cord injury, prostate cancer, bladder cancer, interstitial cystitis, or major depression were excluded. Patient ever received low intensity shockwave or who does not have sex intercourse in recent six months will be excluded.

Measurement of outcomes

Primary outcome: the 4th week and the 8th week change from baseline for IIEF-5 score change from baseline for IIEF-5 score.

Secondary outcomes: Penile Doppler Ultrasound (PDU) at 4th and 8th week , EHS, QoL; AEs

Methodology All patients diagnosed of erectile dysfunction will receive blood sampling of serum testosterone and lipid profile at the beginning of the study. All patients were treated at out-patient clinic. 30 subjects receive LI-ESWT (LM-IASO, Litemed Co., Taiwan) for 6 courses in 3 weeks (0.05mJ/mm2, 3000 pulses) and 30 subjects receive Sham therapy for 3 weeks (the machine turning on but the energy is zero). LI-ESWT is delivered by a probe that was attached to a electrohydraulic unit with a wide-focused shockwave source. The penis is manually stretched, and shockwaves are delivered to the whole penis shaft and penis base. The duration of each ESWT session is about 30 minutes, and comprised 3000 pulses (0.05mJ/mm2), and a frequency of 100/min.

Safety Considerations The peri- and post-treatment adverse events (AEs), including local pain, edema or hematoma were recorded and compared. With consideration of safety issue, any moderate/severe local pain or hematoma would be immediately reported and well inspected.

Follow-up The following parameters are assessed before treatment and weekly during the treatment: IIEF-5 score, EHS, QoL; AEs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 20 ~ 70 year-old man, suffering from ED for over 6 months.
2. 5 ≦ IIEF-5 ≦ 21.

Exclusion Criteria:

1. Patients with penile implant, prior radical prostatectomy, rectal surgery, radiation therapy to the pelvic area, spinal cord injury, prostate cancer, bladder cancer, interstitial cystitis, or major depression.
2. Patient ever received low intensity shockwave or who does not have sex intercourse in recent six months.

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
IIEF-5 score | the 4th week and the 8th week
  the 4th week and the 8th week change from baseline for IIEF-5 score change from baseline for IIEF-5 score.
  The IIEF-5 Questionnaire
  Over the past 6 months:
  1. How do you rate your confidence that you could get and keep an erection? (1-5)
  2. When you had erections with sexual stimulation, how often were your erections hard enough for penetration? (1-5)
  3. During sexual intercourse, how often were you able to maintain your erection after you had penetrated your partner? (1-5)
  4. During sexual intercourse, how difficult was it to maintain your erection to completion of intercourse? (1-5)
  5. When you attempted sexual intercourse, how often was it satisfactory for you? (1-5) Total Score: 1-7: Severe ED 8-11: Moderate ED 12-16: Mild-moderate ED 17-21: Mild ED 22-25: No ED

SECONDARY OUTCOMES:
Penile Doppler Ultrasound (PDU) | the 4th week and the 8th week
  PDU at 4th and 8th week
EHS（Erection Hardness Score） | the 4th week and the 8th week
  EHS at 4th and 8th week EHS score
  How would you rate the hardness of your erection? select one of the following options:
  * 0 - Penis does not enlarge.
  * 1 - Penis is larger, but not hard.
  * 2 - Penis is hard, but not hard enough for penetration.
  * 3 - Penis is hard enough for penetration, but not completely hard.
  * 4 - Penis is completely hard and fully rigid.
QoL: questionnaire | the 4th week and the 8th week
  Quality-of-life questionnaire at 4th and 8th week
  Score 0 (the best) - 6 (the worst)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sokolakis I, Hatzichristodoulou G. Clinical studies on low intensity extracorporeal shockwave therapy for erectile dysfunction: a systematic review and meta-analysis of randomised controlled trials. Int J Impot Res. 2019 May;31(3):177-194. doi: 10.1038/s41443-019-0117-z. Epub 2019 Jan 21. PMID 30664671
- [Result] Campbell JD, Trock BJ, Oppenheim AR, Anusionwu I, Gor RA, Burnett AL. Meta-analysis of randomized controlled trials that assess the efficacy of low-intensity shockwave therapy for the treatment of erectile dysfunction. Ther Adv Urol. 2019 Mar 29;11:1756287219838364. doi: 10.1177/1756287219838364. eCollection 2019 Jan-Dec. PMID 30956690
- [Result] Dong L, Chang D, Zhang X, Li J, Yang F, Tan K, Yang Y, Yong S, Yu X. Effect of Low-Intensity Extracorporeal Shock Wave on the Treatment of Erectile Dysfunction: A Systematic Review and Meta-Analysis. Am J Mens Health. 2019 Mar-Apr;13(2):1557988319846749. doi: 10.1177/1557988319846749. PMID 31027441